CLINICAL TRIAL: NCT01116232
Title: A Pilot Phase II Study of Sirolimus, Tacrolimus, Thymoglobulin and Rituximab as Graft-versus-Host-Disease Prophylaxis in Patients Undergoing Haploidentical and HLA Partially Matched Donor Hematopoietic Cell Transplantation
Brief Title: Sirolimus, Tacrolimus, Thymoglobulin and Rituximab as Graft-versus-Host-Disease Prophylaxis in Patients Undergoing Haploidentical and HLA Partially Matched Donor Hematopoietic Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding.
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Zaid Al-Kadhimi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000671822; P30CA022453 (NIH); U4781s (Other: Genentech); 2009-150 (Other: Barbara Ann Karmanos Cancer Institute); NCT01534767 (obsolete NCT alias)
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Chronic Myeloproliferative Disorders; Graft Versus Host Disease; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: graft versus host disease; accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult T-cell leukemia/lymphoma; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; relapsing chronic myelogenous leukemia; stage I adult T-cell leukemia/lymphoma; stage I chronic lymphocytic leukemia; stage II adult T-cell leukemia/lymphoma; stage II chronic lymphocytic leukemia; stage III adult T-cell leukemia/lymphoma; stage III chronic lymphocytic leukemia; stage IV adult T-cell leukemia/lymphoma; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated hairy cell leukemia; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; cutaneous B-cell non-Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; Waldenstrom macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; stage I adult Burkitt lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage I mantle cell lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III small lymphocytic lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV small lymphocytic lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; intraocular lymphoma; post-transplant lymphoproliferative disorder; chronic eosinophilic leukemia; chronic neutrophilic leukemia; primary myelofibrosis; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable
MeSH Terms: conditions — Myeloproliferative Disorders; Graft vs Host Disease; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Leukemia, Prolymphocytic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, Extranodal NK-T-Cell; Waldenstrom Macroglobulinemia; Lymphoma, B-Cell, Marginal Zone; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Intraocular Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Leukemia, Neutrophilic, Chronic; Primary Myelofibrosis | interventions — Antilymphocyte Serum; Rituximab; Sirolimus; Tacrolimus; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-thymocyte globulin, rituximab, sirolimus, tacrolimus, (Experimental): anti-thymocyte globulin: Infuse the first dose over a minimum of 6 hours, and subsequent doses over a minimum of 4 hours via a 0.22 micron in-line filter
  Rituximab: The total dose chosen for this protocol is 28 mg/kg divided in two doses (14 mg/kg on days -7 and +3). Initial infusion: Start rate of 50 mg/hour;
  For adults, Sirolimus will be administered at 12 mg orally loading dose on day -3, followed by 4 mg orally single morning daily dose (target serum level 3-12 ng/ml by HPLC).
  Tacrolimus will be administered intravenously at a dose of 0.03 mg/kg (ideal body weight) q 24h by continuous infusion starting on Day -3. Intravenous Tacrolimus will be discontinued once the patient starts eating and the drug will then be given orally at a dose of approximately 4 times the intravenous dose.
  Interventions: Biological: anti-thymocyte globulin; Biological: rituximab; Drug: sirolimus; Drug: tacrolimus; Other: laboratory biomarker analysis; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: management of therapy complications; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: anti-thymocyte globulin — Infuse the first dose over a minimum of 6 hours, and subsequent doses over a minimum of 4 hours via a 0.22 micron in-line filter.
Biological: rituximab — The total dose chosen for this protocol is 28 mg/kg divided in two doses (14 mg/kg on days -7 and +3). Initial infusion: Start rate of 50 mg/hour; if there is no reaction, increase the rate by 50 mg/hour increments every 30 minutes, to a maximum rate of 400 mg/hour. Subsequent infusions: If patient did not tolerate initial infusion follow initial infusion guidelines. If patient tolerated initial infusion, start at 100 mg/hour; if there is no reaction, increase the rate by 100 mg/hour increments every 30 minutes, to a maximum rate of 400 mg/hour. Note: If a reaction occurs, slow or stop the infusion. If the reaction abates, restart infusion at 50% of the previous rate.
  In patients who tolerated the Rituximab well in the past, a rapid infusion rate can be used over 90 minutes with 20% of the dose administered in the first 30 minutes and the remaining 80% is given over 60 minutes.
  Other Names: Rituxan®
Drug: sirolimus — For adults, Sirolimus will be administered at 12 mg orally loading dose on day -3, followed by 4 mg orally single morning daily dose (target serum level 3-12 ng/ml by HPLC).
  Other Names: Rapamune®
Drug: tacrolimus — Tacrolimus will be administered intravenously at a dose of 0.03 mg/kg (ideal body weight) q 24h by continuous infusion starting on Day -3. Intravenous Tacrolimus will be discontinued once the patient starts eating and the drug will then be given orally at a dose of approximately 4 times the intravenous dose.
  Other Names: Prograf
Other: laboratory biomarker analysis — laboratory biomarker analysis
Procedure: allogeneic hematopoietic stem cell transplantation — allogeneic hematopoietic stem cell transplantation
Procedure: management of therapy complications — management of therapy complications
Procedure: peripheral blood stem cell transplantation — peripheral blood stem cell transplantation

SUMMARY:
This Phase II clinical trial was designed for patients with hematologic malignancies in need of donor peripheral blood stem cell transplant, and have no HLA matched donor. Therefore It will test the efficacy of combining sirolimus, tacrolimus, antithymocyte globulin, and rituximab in preventing graft versus host disease in transplants from HLA Haploidentical and partially mismatched donors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the incidence and severity of acute graft-vs-host disease (GVHD) in patients with hematologic malignancies undergoing donor peripheral blood stem cell transplantation who are receiving sirolimus, tacrolimus, anti-thymocyte globulin, and rituximab as GVHD prophylaxis.
* Assess time to engraftment absolute neutrophil count (> 0.5 x 10^9/L for 3 consecutive days) and platelet count (> 20 x 10^9/L for 3 consecutive days) in these patients.
* Determine the safety, as defined by serious adverse events and adverse events related to this immunosuppressive regimen, in the first 6 months after treatment.

Secondary

* Assess the incidence of chronic GVHD measured within 2 years after transplantation.
* Assess overall and disease-free survival at 2 years after transplantation.
* Examine the incidence of opportunistic infections including fungal infections, pneumocystis carinii pneumonia, and viral infections (cytomegalovirus, varicella zoster virus, herpes simplex virus, BK virus, Epstein-Barr virus, and post-transplant lymphoproliferative disorder).
* Assess the incidence of thrombotic microangiopathy within 100 days of transplantation.
* Perform immunocorrelative studies, including T-cell, B-cell, NK-cell, regulatory cell, and allo-reactive T-cell measurement studies via flow cytometry, at 30, 60, 90, and 180 days after transplantation.

OUTLINE: Patients receive rituximab IV on days -7 and 3, tacrolimus IV continuously (may switch to orally when the patient is able to eat) and oral sirolimus beginning on day -3, and anti-thymocyte globulin IV over 6 hours on days -3 to -1. Tacrolimus and sirolimus are tapered at the discretion of the treating physician.

All patients also receive a standard transplant-preparative regimen and undergo transplantation on day 0.

Blood samples are collected before the preparative regimen and at 30, 60, 90, and 180 days after transplantation for correlative immunologic studies.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a hematological malignancy, including:

  * Non-Hodgkin lymphoma
  * Hodgkin lymphoma
  * Acute myeloid leukemia or acute lymphoblastic leukemia
  * Myelodysplastic syndrome (treated or untreated)
  * Chronic myelogenous leukemia
  * Multiple myeloma
  * Chronic lymphocytic leukemia
  * Myelofibrosis and other myeloproliferative disorders
* No suitable related HLA-matched or unrelated HLA-matched (8/8 or 7/8 matched) donor
* Available suitable haploidentical or partial-matched unrelated donor (high-resolution molecular HLA typing is mandatory for HLA Class I and II)

  * No more than 4/8 HLA allele or antigen mismatch for a haploidentical-related first-degree family member donor
  * Only 6/8 or 5/8 allele or antigen match for an unrelated donor
* Scheduled to undergo peripheral blood stem cell transplantation

  * Not receiving bone marrow or ex vivo engineered or processed graft (e.g., CD34+ enrichment, T-cell depletion)
* No documented uncontrolled CNS disease

PATIENT CHARACTERISTICS:

* Karnofsky performance status (PS) 70-100%
* ECOG PS 0-2
* Serum bilirubin < 3 times upper limit of normal (ULN)
* ALT and AST < 3 times ULN
* Creatinine clearance > 60 mL/min
* Ejection fraction > 50%
* Forced vital capacity, FEV_1, or DLCO > 50% predicted
* Negative pregnancy test
* Able to cooperate with oral medication intake
* Patients with coronary heart disease (recent myocardial infarctions, angina, cardiac stent, or bypass surgery in the past 6 months) are eligible provided they are cleared with a stress echo or nuclear myocardial perfusions stress test and a cardiology consult
* No ascites
* No HIV positivity
* No active hepatitis B or C virus infection
* No known contraindication to the administration of sirolimus, tacrolimus, anti-thymocyte globulin, or rituximab

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Not on home oxygen

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-08; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Al-Kadhimi, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cancer center clinic.
Groups:
- Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,: anti-thymocyte globulin: Infuse the first dose over a minimum of 6 hours, and subsequent doses over a minimum of 4 hours via a 0.22 micron in-line filter
  Rituximab: The total dose chosen for this protocol is 28 mg/kg divided in two doses (14 mg/kg on days -7 and +3). Initial infusion: Start rate of 50 mg/hour;
  For adults, Sirolimus will be administered at 12 mg orally loading dose on day -3, followed by 4 mg orally single morning daily dose (target serum level 3-12 ng/ml by HPLC).
  Tacrolimus will be administered intravenously at a dose of 0.03 mg/kg (ideal body weight) q 24h by continuous infusion starting on Day -3. Intravenous Tacrolimus will be discontinued once the patient starts eating and the drug will then be given orally at a dose of approximately 4 times the intravenous dose.
  peripheral blood stem cell transplantation
  sirolimus: For adults, will be administered at 12 mg orally loading dose on day -3, follow
Period: Overall Study
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Started | 4
Completed | 0
Not Completed | 4
Not completed — Progressive diease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (2.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Acute Graft-vs-host Disease (GVHD)
Time Frame: During the first six months post transplant
Population: Study terminated due to lack of funding, no analysis was done for this protocol due to the fact that only four patients were accrued, no data was collected.
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

2. Primary Outcome: Time to Engraftment
Time Frame: During the first six months post transplant
Population: as for outcome 1
Groups:
- Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,: Anti-thymocyte globulin infuse the 1st dose, minimum of 6 hrs subsequent doses minimum of 4 hrs via a 0.22 micron in-line filter
  Rituximab, total dose is 28 mg/kg divided in 2 doses (14 mg/kg, days -7 & +3) Initial infusion, start rate 50 mg/hour
  Sirolimus 12 mg orally loading dose on day -3, followed by 4 mg orally single morning daily dose (target serum level 3-12 ng/ml by HPLC).
  Tacrolimus (IV) dose of 0.03 mg/kg (ideal body weight) every 24hr by continuous infusion starting on Day -3, discontinued once the pt. starts eating & the drug will then be given orally at a dose of approximately 4 times the IV dose.
  .
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

3. Primary Outcome: Safety Assessment
Time Frame: During the first six months post transplant
Population: as for outcome 1
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

4. Secondary Outcome: Incidence of Chronic GVHD
Time Frame: Within two years after transplant
Population: as for outcome 1
Groups:
- Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,: anti-thymocyte globulin: Infuse the first dose over a minimum of 6 hours, and subsequent doses over a minimum of 4 hours via a 0.22 micron in-line filter
  Rituximab: The total dose chosen for this protocol is 28 mg/kg divided in two doses (14 mg/kg on days -7 and +3). Initial infusion: Start rate of 50 mg/hour;
  For adults, Sirolimus will be administered at 12 mg orally loading dose on day -3, followed by 4 mg orally single morning daily dose (target serum level 3-12 ng/ml by HPLC).
  Tacrolimus will be administered intravenously at a dose of 0.03 mg/kg (ideal body weight) q 24h by continuous infusion starting on Day -3. Intravenous Tacrolimus will be discontinued once the patient starts eating and the drug will then be given orally at a dose of approximately 4 times the intravenous dose.
  anti-thymocyte globulin: Infuse the first dose over a minimum of 6 hours, and subsequent doses over a minimum of 4 hours via a 0.22 micron in-line filter.
  rituximab: The total dose chosen
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

5. Secondary Outcome: Incidence of Infections Including Cytomegalovirus, Epstein-Barr Virus Reactivation, and Post-transplant Lymphoproliferative Disorder
Time Frame: At one year
Population: as for outcome 1
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

6. Secondary Outcome: Incidence of Thrombotic Microangiopathy
Time Frame: Within 100 days of HCT
Population: as for outcome 1
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall and Disease-free Survival
Time Frame: At 1 year
Population: as for outcome 1
Groups:
- Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,: Anti-thymocyte globulin infuse the 1st dose, minimum of 6 hrs subsequent doses minimum of 4 hrs via a 0.22 micron in-line filter
  Rituximab, total dose is 28 mg/kg divided in 2 doses (14 mg/kg, days -7 & +3) Initial infusion, start rate 50 mg/hour
  Sirolimus 12 mg orally loading dose on day -3, followed by 4 mg orally single morning daily dose (target serum level 3-12 ng/ml by HPLC).
  Tacrolimus (IV) dose of 0.03 mg/kg (ideal body weight) every 24hr by continuous infusion starting on Day -3, discontinued once the pt. starts eating & the drug will then be given orally at a dose of approximately 4 times the IV dose.
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

8. Secondary Outcome: Immunocorrelative Studies Pre- and Periodically Post-transplantation
Time Frame: Using flow cytometry at 30, 60, 90, and 180 days post transplant.
Population: as for outcome 1
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Anti-thymocyte Globulin, Rituximab, Sirolimus, Tacrolimus,
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Study terminated due to lack of funding. No analysis, patient data on this protocol due to the fact that only four patients was able to be accrued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No